CLINICAL TRIAL: NCT03773588
Title: Spatial Entropy and Surgical Pleth Index Guided Closed Loop Target Controlled Infusion (TCI) Total Intravenous Anaesthesia (TIVA) With Propofol
Brief Title: Entropy and Surgical Pleth Index Guided Closed Loop Target Controlled Infusion Total Intravenous Anesthesia With Propofol
Acronym: Closedloop TCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KVG Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Shivakumar M C, MD, Professor and HEAD, Department of Anesthesiologist and critical care medicine, KVG Medical College and Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMCH01
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia Awareness
Keywords: Closed loop; Entropy; Surgical pleth index; Adequacy of Anesthesia; Target controlled infusion
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Intervention Model Description: Device: Closed-Loop propofol TCI with Entropy and SPI Device: Open-Loop propofol by Target Controlled Infusion Drug: propofol
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Closed-Loop propofol Target control infusion (Active Comparator): Closed loop target controlled infusion(TCI) TIVA with propofol using BD TCI pumps guided by entropy and SPI
  Interventions: Device: Closed-Loop propofol Target controlled infusion by Entropy and SPI
- Open-loop propofol target control infusion (Active Comparator): Open-loop target controlled infusion of propofol using BD TCI pumps based on Schnider effect site algorithm
  Interventions: Device: Open-loop propofol target controlled infusion

INTERVENTIONS:
Device: Closed-Loop propofol Target controlled infusion by Entropy and SPI — Closed loop target infusion of propofol using BD TCI pumps guided by entropy and Surgical pleth index
  Other Names: Closed-loop propofol Target controlled infusion
  Arms: Closed-Loop propofol Target control infusion
Device: Open-loop propofol target controlled infusion — Propofol target controlled infusion using Schnider algorithm to determine effect site concentration
  Other Names: Open-loop propofol TCI
  Arms: Open-loop propofol target control infusion

SUMMARY:
Closed-loop infusion system for target controlled infusion of propofol by using TCI pump designed by BD Technology. (Germany) guided with entropy and surgical pleth index (GE) will not only prevent awareness from Anesthesia but also optimise the dose anesthetic agents based on feedback from adequacy of Anesthesia monitoring. Which not only reduces Anesthesia agents but also enhances recovery from Anesthesia. Innovation using TCI combined with closed-loop controlled intravenous anesthesia under the guide of Entropy.In this study we performed a randomized, controlled, study to compare closed-loop control and open-loop control of propofol by using the Entropy and SPI guided closed-loop infusion system.

DETAILED DESCRIPTION:
Monitoring of Adequacy of Anesthesia using Entropy and Surgical pleth index to guide total intravenous anesthesia is more effective to maintain depth of anesthesia compared with target controlled infusion with open systems, it is unclear what driver and variables to achieve this goal be more physiological; in the literature doesn´t exist studies showing that the closed-loop system for hypnotic is better than the controlled algorithm based pharmacokinetic models and open loop system (target controlled infusion-TCI) to maintain anesthetic depth. Thus, a system was designed for intravenous anesthesia in closed loop for propofol as hypnotic based on neuromonitoring with Entropy and surgical pleth index as adequacy of Anesthesia depth.

The purpose of this study is to determine the therapeutic effectiveness of a closed loop TCI for administration of intravenous anesthesia using adequacy of anesthesia monitoring to maintain a depth of anesthesia compared to an open loop system TCI.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Scheduled for noncardiac surgery elective low-risk or intermediate risk. -Expected surgery time greater than 1 hour
* Procedure requiring general anesthesia
* Classification of the American Society of Anesthesiologists (ASA) as I,II, lll

Exclusion Criteria:

* Pregnant women
* Surgery scheduled urgent or emergency
* Personal history of allergy to eggs or any other part of propofol
* Personal history of abnormalities or congenital or acquired cognitive sequels: infantile cerebral palsy, Down syndrome, cerebral ischemic disease, traumatic brain injury, brain tumor, autism.
* Chronic use of benzodiazepines or antipsychotics
* A patient who does not consent to participate in the study prior to surgery or before randomization
* Need for anesthetic or analgesic blockade before surgery peripheral nerve

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-01-10 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Adequacy of anesthesia | 1 day
  Difference in therapeutic effectiveness determined by the time in state suitable anesthetic depth. The proper anesthetic depth is defined as the efficacy to maintain a Spatial entropy in the range of 40 - 60 during a surgery.
Time taken for recovery from Anesthesia | 1 day
  Total time taken for recovery after stopping of infusion

SECONDARY OUTCOMES:
Total consumption of propofol | 1 day
  Total consumption of propofol during surgery
Number of hypotension events | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Subbaih institute of medical sciences, Shimoga, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided